CLINICAL TRIAL: NCT01525784
Title: Prospective Short and Long Term Follow up of Pediatric Diabetes Mellitus Patients Receiving RT-CGMS as Part of National Clinical Care
Brief Title: Affect of RT-CGMS as Part of Clinical Care in Type 1 Diabetes Mellitus Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Soroka University Medical Center (Other); Wolfson Medical Center (Other Government); The Chaim Sheba Medical Center (Other); Kaplan Medical Center (Other)
Responsible Party: Principal Investigator, Assaf Harofeh MC, Dr. Marianna Rachmiel, Assaf Haroffeh Medical Center, Assaf-Harofeh Medical Center
Other Study IDs: 88\11
Record Dates: First submitted 2011-11-03; First posted 2012-02-03 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Hypoglycemia; Type 1 Diabetes Mellitus
Keywords: rtCGMS; glycemic control; type 1 diabetes mellitus; youth
MeSH Terms: conditions — Hypoglycemia; Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Rt-CGMS: Using Rt-CGMS, approved by ministry of health as part f clinical care
- Control: Not approved or suggested for RtCGMS. Other acceptabl means of therapy

SUMMARY:
The incidence of Type 1 Diabetes Mellitus is increasing annually, in all pediatric age groups, especially among infants and toddlers.However, only 30% of diabetic children manage to achieve and maintain glycated hemoglobin A1c (HbA1c) levels below 8%, although most are treated by intensive insulin therapy.Recently, devices for real-time continuous glucose monitoring (RT-CGMS) have been introduced to aid self management of glycemic control. These devices enable the patients to see the interstitial glucose levels continuously, the trends of decrement and increment, and to have alarms prior to a severe hypoglycemic episode .

The RT-CGMS was approved in Israel for routine usage in the pediatric population, 0-18 years in 2011, indicated for those with recurrent hypoglycemic episodes. So, the aim of the investigators study is to examine prospectively the short and long term effect of the RT-CGMS routine usage, in daily routine life of the diabetic child.

DETAILED DESCRIPTION:
The incidence of Type 1 Diabetes Mellitus is increasing annually, in all pediatric age groups, especially among infants and toddlers.

However, only 30% of diabetic children manage to achieve and maintain glycated hemoglobin A1c (HbA1c) levels below 8%, although most are treated by intensive insulin therapy by multiple daily injections (MDI) or by subcutaneous continuous insulin infusion (SCII). The presence of high HbA1c levels increase the probability for long term complications of diabetes, as retinopathy, nephropathy and neuropathy.

This failure is attributed to multiple reasons; irregular meals, unpredictable physical activity, behavioral difficulties, refusal to accept the diabetes and maintain the required lifestyle, resistance to insulin, but , most of all fear of hypoglycemia and hypoglycemia unawareness . Further more, recurrent hypoglycemic episodes under the age of 6 years old may cause neurocognitive permanent damage.

Recently, devices for real-time continuous glucose monitoring (RT-CGMS) have been introduced to aid self management of glycemic control. These devices enable the patients to see the interstitial glucose levels continuously, the trends of decrement and increment, and to have alarms prior to a severe hypoglycemic episode .

Only few studies were performed in the pediatric population. One showed a decrement of 0.27% in HbA1c after 1 month and the other a 1 % decrement in 50% of study population after 3 months, but in the adult population. A study performed in the minority group of well controlled diabetic patients (HA1c<7.5%) demonstrated an increment of 1.56 hours per day of normoglycemia, and less time spent an hypoglycemia among those using RT-CGMS for 26 weeks.

However, those studies were performed in chosen groups and motivated patients, in a state of research with multiple clinic visits and reminders. Those studies do not always reflect the real life benefit of the equipment and its best usage method.

The RT-CGMS was approved in Israel for routine usage in the pediatric population, 0-18 years in 2011, indicated for those with recurrent hypoglycemic episodes.

The aim of our study

* to examine prospectively the short and long term effect of the RT-CGMS routine usage, in daily routine life of the diabetic toddler, child and adolescent on glycemic control, frequency of day time and nocturnal hypoglycemia and quality of life not under a research template.
* to identify the characteristics of those patients who will benefit most of the RT-CGMS routine usage.
* to identify the characteristics of those patients who will not benefit, but will even worsen of the RT-CGMS routine usage

Study design:

This is a prospective multicenter case-control cohort study. We will follow prospectively all patients receiving RT-CGMS as part of their routine management, for a period of 2 years, in five centers of pediatric diabetes care in Israel.

All participants will receive similar guidance and instructions prior to RT-CGMS usage.

All clinic visits, at intervals of 3 months or more will be recorded, including data regarding weight, height, insertion sites, blood glucose average measurements, CGMS measurements and variability, frequency of hypoglycemia, time spent in normoglycemia and HbA1c.

Quality of Life and Anxiety questionnaires will be filled bi-annually.

ELIGIBILITY:
Inclusion Criteria:

* Age 1-18 years
* Type 1 Diabetes Mellitus

Exclusion Criteria:

* Refusal to participate

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All patients recieving CGMS for treatment group and those without RTCGMS but all other management, for control group.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-02; Primary Completion 2014-01 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
to examine prospectively frequency of hypoglycemia | 3 years

SECONDARY OUTCOMES:
to assess the effect of rt-cgms on quality of life of children and parents | 3 years
To examine prosectively the effect of rt-cgms on glycemic control | 3 years
  to follow the effect of rt-cgms on hba1c and on bg average and complications

CONTACTS AND LOCATIONS:
Overall Officials: Marianna rachmiel, md, Principal Investigator — Assaf Haroffeh Medical Center
Locations (4):
- Israel (4):
  - Soroka University Medical Center, Beersheba
  - Wolfson Medical Center, Holon
  - Sheba Medical Center, Tel Aviv
  - Assaf harofeh Medical Center, Ẕerifin

REFERENCES:
- [Derived] Rachmiel M, Landau Z, Boaz M, Mazor Aronovitch K, Loewenthal N, Ben-Ami M, Levy-Shraga Y, Modan-Moses D, Haim A, Abiri S, Pinhas-Hamiel O. The use of continuous glucose monitoring systems in a pediatric population with type 1 diabetes mellitus in real-life settings: the AWeSoMe Study Group experience. Acta Diabetol. 2015 Apr;52(2):323-9. doi: 10.1007/s00592-014-0643-6. Epub 2014 Sep 16. PMID 25223531